CLINICAL TRIAL: NCT02268773
Title: A Randomised, Two-period, Cross-over Trial to Compare the Effects of Acetylsalicylic Acid (75 mg/Day) With the Combination of Acetylsalicylic Acid (25 mg) + Modified-release Dipyridamole (200 mg) (bd) on Serum Thromboxane B2 Formation and Platelet Aggregation in Healthy Volunteers
Brief Title: Effects of Acetylsalicylic Acid Compared With the Combination of Acetylsalicylic Acid + Modified-release Dipyridamole on Serum Thromboxane B2 Formation and Platelet Aggregation in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 9.130
Record Dates: First submitted 2014-10-17; First posted 2014-10-20 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Aspirin, Dipyridamole Drug Combination; Aspirin

ARMS (2):
- Acetylsalicylic acid low dose with Asasantin® (Experimental)
  Interventions: Drug: Asasantin®; Drug: Acetylsalicylic acid low dose
- Acetylsalicylic acid high dose (Active Comparator)
  Interventions: Drug: Acetylsalicylic acid high dose

INTERVENTIONS:
Drug: Asasantin®
  Other Names: modified-release dipyridamole
  Arms: Acetylsalicylic acid low dose with Asasantin®
Drug: Acetylsalicylic acid low dose
  Arms: Acetylsalicylic acid low dose with Asasantin®
Drug: Acetylsalicylic acid high dose
  Arms: Acetylsalicylic acid high dose

SUMMARY:
To compare the combination of acetylsalicylic acid (25 mg) + modified-release dipyridamole (200 mg) bd versus acetylsalicylic acid (75 mg dispersible tablet once daily) in its effect on inhibition of thromboxane B2 formation

ELIGIBILITY:
Inclusion Criteria:

* Male or female healthy volunteers aged 20 to 50 years
* Clinically normal medical history
* Clinically normal findings on physical examination
* Capable of comprehending and communicating effectively with the investigator and staff and of providing informed consent
* Willing to give informed consent prior to participation in the trial (i.e. prior to any trial-specific procedures)

Exclusion Criteria:

* Any clinically significant disease. (A significant disease is defined as a disease which in the opinion of the investigator may either put the subject at risk because of participation in the study or a disease which may influence the results of the study or the subject's ability to participate in the study)
* Clinically significant abnormal baseline haematology, blood chemistry or urinalysis findings
* Serum glutamate-oxaloacetate transferase (SGOT) or serum glutamate-pyruvate transferase (SGPT) > 80 IU/L, bilirubin > 34 µmol/L or creatinine > 176 µmol/L regardless of clinical condition. Repeat laboratory evaluation will not be conducted in these subjects
* Use of dipyridamole, aspirin or any non-steroidal anti-inflammatory agent (NSAID) during the previous two weeks
* Active peptic ulceration or history of peptic ulcer disease
* Known history of or suspected hypersensitivity to dipyridamole, aspirin, any NSAID or any other component of the test drugs
* History of any bleeding disorders
* History of cerebral haemorrhage
* Resting, seated blood pressure less than 90/60 mmHg
* Participation in any drug clinical trial within sixteen weeks prior to the start of the trial
* Any indication of current or previous abuse of alcohol, solvents or drugs
* Any chronic illness
* Asthma
* Requirement for any other medication one month before or during the study
* Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception (e.g. oral contraceptives, intrauterine devices or surgically sterile) were to be excluded
* Previous participation in the randomisation phase of this clinical trial

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2000-01; Primary Completion 2000-05 (Actual)

PRIMARY OUTCOMES:
Absolute serum thromboxane B2 level | At day 3 after start of drug administration

SECONDARY OUTCOMES:
Change in platelet aggregation | At day 3 after start of drug administration
  measured ex-vivo
Change in time course of inhibition of serum thromboxane B2 | Pre-dose, up to day 14 after start of drug administration
Change in time course of inhibition of platelet aggregation | Pre-dose, up to day 14 after start of drug administration
Changes from baseline in vital signs | Pre-dose, up to 14 days after first drug administration
  systolic and diastolic blood pressure, pulse rate
Changes from baseline in laboratory tests | Pre-dose, up to 14 days after first drug administration
Changes from baseline in physical examination | Pre-dose, up to 14 days after first drug administration
Changes from baseline in 12-lead ECG | Pre-dose, up to 14 days after first drug administration
Number of patients with adverse events | Up to 14 days after start of drug administration